CLINICAL TRIAL: NCT01941316
Title: Phase 1b/II Trial of Carfilzomib With Irinotecan in Irinotecan-Sensitive Malignancies (Phase Ib) and Small Cell Lung Cancer Patients (Phase II) Who Have Progressed on Prior Platinum-based Chemotherapy
Brief Title: Study of Carfilzomib With Irinotecan in Irinotecan-Sensitive Malignancies and Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research and Biostatistics Clinical Trials Consortium (Network)
Collaborators: Lucille P. Markey Cancer Center at University of Kentucky (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRAB CTC 11-001; CAR-IST-553 (Other: Onyx Pharmaceuticals)
Record Dates: First submitted 2013-08-19; First posted 2013-09-13 (Estimated); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Small Cell Lung Carcinoma; Non Small Cell Lung Carcinoma; Irinotecan Sensitive Cancers
Keywords: Carfilzomib; Irinotecan; Small Cell Lung Cancer; Non Small Cell Lung Cancer; Ovarian Cancer; Gastric Cancer; Esophageal Cancer; Cervical Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms | interventions — carfilzomib; Irinotecan

STUDY DESIGN:
Intervention Model Description: A total of 16 patients were enrolled to the Phase 1b run-in at 3 different dosing levels:
  4 patients into Dosing Level 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan
  9 patients into Dosing Level 2: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan
  3 patients into Dosing Level 3: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan
  A total of 62 patients were enrolled into the Phase 2 trial. The Phase 2 component is a single-arm component, with participants stratified into two groups:
  37 platinum-sensitive
  25 platinum-refractory
  Enrollment was not sequential, as all participants in the Phase 2 component were different individuals than the participants enrolled into the Phase 1b component.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase II (Experimental): Phase II: Stratified, single arm trial using a starting dose of 20/36 mg/m^2 of carfilzomib and 125 mg/m^2 of irinotecan, in small cell lung cancer patients who have relapsed on a prior platinum regimen.
  Stratification for phase II component:
  1. Platinum sensitive disease: initial response to platinum-based chemotherapy with progression > 90 days after last treatment.
  2. Platinum refractory disease: No response to platinum-based chemotherapy or progression within 90 days of completing platinum-based therapy. Subjects that progressed during or within one month of completion of platinum-based chemotherapy will be excluded.
  Interventions: Drug: Carfilzomib; Drug: Irinotecan
- Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (Experimental): Cohort 1 of Phase Ib run-in to determine maximum tolerated dose (MTD) of Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
  Cohort 1 used a starting dose of 20/27 mg/m^2 of carfilzomib in combination with 125 mg/m^2 of irinotecan.
  Interventions: Drug: Carfilzomib; Drug: Irinotecan
- Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (Experimental): Cohort 2 of Phase Ib run-in to determine maximum tolerated dose (MTD) of Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
  Cohort 2 used a starting dose of 20/36 mg/m^2 of carfilzomib in combination with 125 mg/m^2 of irinotecan.
  Interventions: Drug: Carfilzomib; Drug: Irinotecan
- Phase Ib Cohort 1: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (Experimental): Cohort 3 of Phase Ib run-in to determine maximum tolerated dose (MTD) of Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
  Cohort 3 used a starting dose of 20/45 mg/m^2 of carfilzomib in combination with 125 mg/m^2 of irinotecan.
  Interventions: Drug: Carfilzomib; Drug: Irinotecan

INTERVENTIONS:
Drug: Carfilzomib — 20/36 * mg/m^2 stepped up dosing, IV infusion (over 30 min), on days 1, 2, 8, 9, 15 and 16 of each 28 day cycle. Number of cycles: 6, or until progression, or unacceptable toxicity, or treatment delay for any reason greater than 3 weeks.
  Other Names: Kyprolis
Drug: Irinotecan — 125 mg/m^2, IV infusion (over 90 min), on days 1, 8, 15 of each 28 day cycle. Number of cycles: 6, or until progression, or unacceptable toxicity, or treatment delay for any reason greater than 3 weeks.
  Other Names: Camptosar; Campto

SUMMARY:
The purpose of this study is to determine a well-tolerated dose of Carfilzomib in combination with Irinotecan (Phase 1b portion of the study) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers and to assess the 6 month survival of relapsed small cell lung cancer patients treated with this combination therapy. **The Phase 1b portion of the study is now complete**.

Phase 2 portion of the study. The safest, maximally tolerated dose established as established in Phase 1 for Phase 2 is as follows -- Carfilzomib will be provided at 20/36 mg/m^2 with Irinotecan dosed at 125 mg/m^2. The purpose of the Phase 2 portion of the study is to assess 6 month survival of relapsed small cell lung cancer ins subjects treated with this combination therapy.

DETAILED DESCRIPTION:
Small cell lung cancer accounts for approximately 15% of all lung cancer diagnoses in the United States (US), with 60-80% response rates to platinum-based chemotherapy in extensive disease. Despite its sensitivity to chemotherapy, small cell lung cancer is characterized by its tendency to spread to other locations in the body such as the bloodstream and other organs such as the liver. Currently, the only FDA-approved second-line therapies are oral and parenteral topotecan, although irinotecan is also commonly used in primary and relapsed disease. Novel combination therapies are desperately needed in this disease. in order to improve survival.

Carfilzomib (also known as Kyprolis) is an anti-cancer drug classified as a selective proteasome inhibitor. Proteasome inhibition affects the levels of numerous cell cycle control proteins, apoptosis (i.e., cell death), cell adhesion, angiogenesis, and chemoresistance proteins. Chemically, it is similar to epoxomicin.

Carfilzomib and other proteasome inhibitors interrupt cellular pathways integral to the survival of small cell lung cancer, namely the apoptotic pathway involving activated Nuclear Factor-kB (referenced as NF-kB). NF-kB activates the transcription of anti-apoptotic and proliferation genes, mediating tumor cell survival in response to cytotoxic stress thus resulting in chemoresistance, a common problem in small cell lung cancer. Carfilzomib prevents the breakdown of IkappaB (referenced as IkB), a protein which inhibits NF-kB, controls levels of the anti-apoptotic gene Bcl-2 and the tumor suppressor p53. Overexpression of Bcl-2, a key mediator of resistance to apoptosis following chemotherapy, which is an important problem in small cell lung cancer.

In this trial, Carfilzomib is combined with Irinotecan. Irinotecan, a camptothecins, inhibits topoisomerase I, thought to be important in the growth and spread of cancer. As a class, camptothecins have shown efficacy in small cell lung cancer in a variety of settings.

Topoisomerase-1 is thought to cause apoptosis via mechanisms other than NF-kB, adding to the potential synergy of these compounds. In addition, topoisomerase-1 is overexpressed in the majority of subjects with small cell lung cancer and decreased degradation of this enzyme is expected to lead to further enhancement of this mechanism of apoptosis

The pivotal phase III study which led to FDA approval of topotecan in relapsed small cell lung cancer was by Von Pawel et al, and included 211 subjects with sensitive (> 60 days since prior therapy) relapse and randomized them to either topotecan (107 subjects) daily for 5 days or to cyclophosphamide, doxorubicin, and vincristine (CAV), each given every 21 days. Topotecan showed no significant improvement in the median time to progression (13.3 weeks vs.12.3 weeks, p=0.552) or median survival (25 weeks vs. 24.7 weeks, p=0.795), however, subjects treated with topotecan had improvement in cancer-related symptoms (dyspnea, hoarseness, anorexia, and fatigue) as well as hematologic toxicity. Irinotecan, has established activity in small cell lung cancer, as well as non-small cell lung cancer, colorectal cancer and ovarian cancer.

In this Phase 2 study patients will be treated with the Maximum Tolerated Dose (MTD) of Carfilzomib 20/36 mg/m^2 as stepped up dosing determined in Phase 1b and 125mg/m^2 of Irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically-confirmed diagnosis of progressive or recurrent malignancy as follows:
* Phase II: extensive stage small cell lung cancer with progression or recurrence after exactly one platinum-containing regimen. Patients who progressed during or within one month of completing platinum-based chemotherapy will be excluded. Patients who received primary curative chemoradiation therapy for limited disease, but who recur within the primary tumor site, previously radiated field or with distant metastases are also allowed to participate. Patients who have clinical evidence of recurrent small cell lung cancer do not require a confirmatory biopsy to be eligible for this trial. Prior irinotecan is not allowed.
* Patients must have measurable disease per RECIST criteria 1.1 performed within 28 days prior to enrollment. All other required tests to assess non-measurable disease must be performed within 42 days prior to enrollment.
* Patients with known brain metastases are eligible only if he/she has been treated for brain metastasis, are asymptomatic after treatment, have a stable CT or MRI of the brain within 28 days of enrollment and are not receiving corticosteroid therapy to control symptoms from brain metastasis. Only a non-enzyme inducing anticonvulsant (e.g., Keppra) will be permitted for those patients requiring anticonvulsants. (Topical and/or inhaled steroids are allowed.)
* Patients may have received previous radiation therapy, but it must have been completed at least 21 days prior to enrollment and the patient should have recovered from all associated toxicities. Measurable or non-measurable disease must be present outside the previous radiation field or a new lesion inside the radiation port must be present.
* Patients may have received prior surgery provided that at least 28 days have elapsed since major surgery (thoracic or other major surgeries) and the patient has recovered from all associated toxicities. Patients must have disease outside of the previous surgical resection area or a new lesion must be present.
* Patients must have a serum creatinine ≤ the institutional upper limit of normal OR a creatinine clearance ≥ 60 cc/min, measured or calculated (Cockcroft-Gault formula), obtained within 14 days prior to registration.
* Patients must have adequate hepatic function as documented by a bilirubin ≤ 2 x the institutional upper limit of normal, an alkaline phosphatase ≤ 2 x the institutional upper limit of normal, and an Serum Glutamate Oxaloacetic Transaminase (SGOT) and Serum Glutamate Pyruvate Transaminase (SGPT) ≤ 2 x the institutional upper limit of normal all obtained within 14 days prior to enrollment.
* Patients must have an Absolute Neutrophil Count (ANC) ≥ 1,500/μl and a platelet count ≥ 100,000/μl obtained within 14 days prior to registration.
* Patients must be 18 years of age or older.
* Patients must have a Zubrod Performance Status as follows:

  1. Phase Ib: 0 or 1
  2. Phase II: 0, 1 or 2
* Patients must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use an effective contraceptive method (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Male subjects must agree to practice contraception.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* No prior irinotecan or carfilzomib
* Must not have leptomeningeal metastases.
* Must be no anticipated need for concurrent radiation therapy during protocol treatment.
* Subjects that progressed during or within one month of completion of first-line platinum-based chemotherapy will be excluded.
* Patients must not be pregnant or lactating females.
* Must have had no major surgery within 28 days prior to enrollment.
* Must not have acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrollment.
* Must not have any known human immunodeficiency virus infection.
* Must not have known active or clinically significant hepatitis A, B or C infection.
* Must not have had any unstable angina or myocardial infarction within 4 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
* Must not have any uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment.
* Must not have any evidence of other clinically active cancer and have no history of prior malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal glands or pancreas.
* Must not have any significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to enrollment.
* Must not have any known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
* Must have no contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
* Must not have any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-11; Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Arnold, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (8):
- United States (8):
  - Cancer Treatment Centers of America, Western Regional Medical Center, Goodyear, Arizona
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - Providence Portland Medical Center | Earle A. Chiles Research Institute, Portland, Oregon
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Virginia Mason Cancer Institute, Seattle, Washington
  - Aurora Research Institute | Aurora Cancer Care, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m2 Irinotecan: Cohort 1 of Phase Ib run-in to determine maximum tolerated dose (MTD) of Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
  Cohort 1 used a starting dose of 20/27 mg/m^2 of carfilzomib in combination with 125 mg/m^2 of irinotecan.
- Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m2 Irinotecan: Cohort 2 of Phase Ib run-in to determine maximum tolerated dose (MTD) of Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
  Cohort 2 used a starting dose of 20/36 mg/m^2 of carfilzomib in combination with 125 mg/m^2 of irinotecan.
- Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m2 Irinotecan: Cohort 3 of Phase Ib run-in to determine maximum tolerated dose (MTD) of Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
  Cohort 3 used a starting dose of 20/45 mg/m^2 of carfilzomib in combination with 125 mg/m^2 of irinotecan.
- Phase II: Trial of Carfilzomib With Irinotecan, SCLC Subjects: Phase II: Stratified, single arm trial, starting dose of 20/36 mg/m2 of carfilzomib and 125 mg/m2 of irinotecan, small cell lung cancer patients who relapsed on a prior platinum regimen.
  Stratification:
  Platinum sensitive disease: initial response to platinum-based chemotherapy with progression > 90 days after last treatment.
  Platinum refractory disease: No response to platinum-based chemotherapy or progression within 90 days of completing platinum-based therapy. Subjects who progressed within 1 month of completed platinum-based chemotherapy were excluded.
  Carfilzomib: 20/36 mg/m2 stepped up dosing, IV infusion (30 min), days 1, 2, 8, 9, 15 and 16 of each 28 day cycle. # cycles: 6, until progression, or unacceptable toxicity, or treatment delay for any reason greater than 3 weeks.
  Irinotecan: 125 mg/m2, IV infusion (90 min), days 1, 8, 15 of each 28 day cycle. # cycles: 6, until progression, or unacceptable toxicity, or treatment delay for any reason greater than 3 weeks.
Period: Overall Study
Arm/Group | Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m2 Irinotecan | Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m2 Irinotecan | Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m2 Irinotecan | Phase II: Trial of Carfilzomib With Irinotecan, SCLC Subjects
Started | 4 | 9 | 3 | 62
Completed | 1 | 0 | 0 | 7
Not Completed | 3 | 9 | 3 | 55
Not completed — Adverse Event | 0 | 1 | 0 | 7
Not completed — Progressive Disease | 3 | 6 | 2 | 29
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 8
Not completed — Death | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 3
Not completed — Intercurrent illness | 0 | 0 | 0 | 1
Not completed — Other, not specified | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan: Cohort 3 of Phase Ib run-in to determine maximum tolerated dose (MTD) of Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
  Cohort 3 used a starting dose of 20/45 mg/m^2 of carfilzomib in combination with 125 mg/m^2 of irinotecan.
- Total: Total of all reporting groups
Arm/Group | Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase II | Total
Number analyzed (Participants) | 4 | 9 | 3 | 62 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 1 | 26 | 34
  >=65 years | 0 | 6 | 2 | 36 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 34 | 42
  Male | 1 | 5 | 2 | 28 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 3
  White | 3 | 9 | 3 | 59 | 74
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Maximum Tolerated Dose
Description: Maximum tolerated dose of Carfilzomib in combination with Irinotecan in subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers.
Time Frame: 28 Days
Population: Subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers. Subjects were given Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in a standard 3+3 dose-finding design.
Measure: Number; unit: mg/m^2 Carfilzomib
Groups:
- Phase 1b: All Patients Enrolled for MTD Determination of Carfilzomib With Irinotecan: 16 total subjects with relapsed small and non-small cell lung cancer or other irinotecan-sensitive cancers. Subjects were given Carfilzomib (Day 1,2,8,9, 15, and 16) in combination with Irinotecan (Days 1, 8, 15) in a standard 3+3 dose-finding design.
Arm/Group | Phase 1b: All Patients Enrolled for MTD Determination of Carfilzomib With Irinotecan
Number analyzed (Participants) | 16
mg/m^2 Carfilzomib
  MTD for Cycle 1 Day 1 and Day 2 doses | 20
  MTD for all doses after Cycle 1 Days 1 and 2 | 36

2. Primary Outcome: Phase II: Overall Survival Rate at 6 Months
Description: Estimate of 6-month overall survival (OS) rate of relapsed small cell lung cancer patients treated with Carfilzomib in combination with Irinotecan.
  The survival function was estimated using the Kaplan-Meier method, with overall survival defined as time from enrollment until death. Patients with no date of death were censored at the time of last contact.
Time Frame: up to 6 Months
Population: A total of 62 eligible relapsed small cell lung cancer patients treated with Carfilzomib in combination with Irinotecan.
Measure: Number (95% Confidence Interval); unit: Proportion with 6-month OS by KM
Groups:
- Platinum Sensitive Disease: Initial response to platinum-based chemotherapy with progression > 90 days after last treatment.
- Platinum Refractory Disease: No response to platinum-based chemotherapy or progression within 90 days of completing platinum-based therapy. Subjects that progressed during or within one month of completion of platinum-based chemotherapy will be excluded.
Arm/Group | Platinum Sensitive Disease | Platinum Refractory Disease
Number analyzed (Participants) | 37 | 25
Proportion with 6-month OS by KM | 0.59 [0.41 to 0.73] | 0.54 [0.33 to 0.71]

3. Secondary Outcome: Overall Response Rate
Description: Rate of overall response of relapsed small cell lung cancer patients treated with Carfilzomib in combination with Irinotecan.
  Responses were evaluated by the criteria defined in RECIST v1.1. Patients were categorized at each response assessment as having one of the following:
  complete response (CR) partial response (PR) stable disease (SD) progressive disease (PD) not assessable (NA)
  Overall response rate is defined as the proportion of patients achieving a best response of PR or better while on study; in other words, the proportion of patients achieving a CR or PR while on study.
Time Frame: From enrollment until the earliest out of date of discontinuation from study or death
Population: Relapsed small cell lung cancer patients treated with Carfilzomib in combination with Irinotecan.
Measure: Number; unit: proportion of patients
Groups:
- Phase II: Platinum Sensitive Disease: Initial response to platinum-based chemotherapy with progression > 90 days after last treatment.
- Phase II: Platinum Refractory Disease: No response to platinum-based chemotherapy or progression within 90 days of completing platinum-based therapy. Subjects who progressed within 1 month of completed platinum-based chemotherapy were excluded.
Arm/Group | Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase II: Platinum Sensitive Disease | Phase II: Platinum Refractory Disease
Number analyzed (Participants) | 4 | 9 | 3 | 37 | 25
proportion of patients | 0.250 | 0.111 | 0.333 | 0.216 | 0.125

4. Secondary Outcome: Phase II: Progression-Free Survival Rate at 6 Months
Description: Estimate of 6-month progression-free survival (PFS) rate of relapsed small cell lung cancer patients treated with Carfilzomib in combination with Irinotecan.
  The survival function was estimated using the Kaplan-Meier method, with progression-free survival defined as time from enrollment until disease progression or death. Patients with no date of death and no date of disease progression were censored at the time of last contact.
Time Frame: up to 6 months
Population: A total of 62 eligible relapsed small cell lung cancer patients treated with Carfilzomib in combination with Irinotecan.
Measure: Number (95% Confidence Interval); unit: Proportion with 6-month PFS by KM
Arm/Group | Platinum Sensitive Disease | Platinum Refractory Disease
Number analyzed (Participants) | 37 | 25
Proportion with 6-month PFS by KM | 0.32 [0.18 to 0.47] | 0.12 [0.03 to 0.28]

5. Secondary Outcome: Phase Ib: Dose Limiting Toxicities
Description: Number of Dose Limiting Toxicity (DLT) adverse events related to Carfilzomib in combination with Irinotecan administration. Subjects were evaluated for toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) of version 4.0.
  A DLT is defined as any of the treatment emergent toxicities with attribution to one or more of the study drugs that occur during Cycle 1.
  Non-hematologic:
  * ≥ Grade 2 neuropathy with pain
  * ≥ Any Grade 3 or 4 toxicity (excluding nausea, vomiting, diarrhea or grade 3 fatigue)
  * ≥ Grade 3 nausea, vomiting, or diarrhea lasting > 7 days despite maximal antiemetic/antidiarrheal therapy
  * ≥ Grade 4 fatigue lasting for ≥ 7 days
  Hematologic:
  Grade 4 neutropenia lasting for ≥ 7 days, Febrile neutropenia, Grade 4 thrombocytopenia lasting ≥ 7 days despite dose delay, Grade 3-4 thrombocytopenia associated with bleeding
Time Frame: up to 6 months
Population: as for outcome 1
Measure: Number; unit: Dose Limiting Toxicities
Arm/Group | Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan
Number analyzed (Participants) | 4 | 9 | 3
Dose Limiting Toxicities
  Dehydration | 0 | 1 | 1
  Diarrhea | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From enrollment until the earliest out of date of study completion, discontinuation from study, or death, an average of 3 months
Arm/Group | Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan | Phase II
All-Cause Mortality (participants affected / at risk) | 2/4 | 5/9 | 1/3 | 51/62
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/9 | 1/3 | 31/62
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 3/3 | 60/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (N=4) | Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (N=9) | Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (N=3) | Phase II (N=62)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 13
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1
Hepatobiliary disorders- Other (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 10
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neoplasms, all (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
RLNP (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Lower GI hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Sudden death NOS (General disorders) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 3
Sepsis (Infections and infestations) | 0 | 0 | 0 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Cohort 1: 20/27 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (N=4) | Phase Ib Cohort 2: 20/36 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (N=9) | Phase Ib Cohort 3: 20/45 mg/m^2 Carfilzomib, 125 mg/m^2 Irinotecan (N=3) | Phase II (N=62)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 24
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac disorder - Other (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1 | 8
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 6
Diarrhea (Gastrointestinal disorders) | 2 | 7 | 2 | 40
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GERD (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 2 | 27
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 6
GI disorders - Other (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 3 | 41
Infusion related reaction (General disorders) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
ALT increased (Investigations) | 1 | 0 | 0 | 5
AST increased (Investigations) | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 15
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 19
Platelet count decreased (Investigations) | 1 | 1 | 2 | 18
Weight loss (Investigations) | 0 | 0 | 1 | 0
White blood cell decreased (Investigations) | 1 | 1 | 1 | 17
Investigations - Other (Investigations) | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 23
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Sinus pain (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 6
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal/urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin/subq tissue ds - Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 4
Hypotension (Vascular disorders) | 0 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT01941316/Prot_SAP_000.pdf